CLINICAL TRIAL: NCT01091116
Title: Intra-articular Treatment With MEN16132 in Patients With Symptomatic Primary Osteoarthritis of the Knee: A Randomized, Multi-centre, Double Blind, Placebo Controlled, Five Parallel Group, Dose Finding Study
Brief Title: A Locally Injected Bradykinin Antagonist for TReatment of OSteoarthritiS
Acronym: ALBATROSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BKOS-02; 2009-014918-99 (EudraCT Number)
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Injections, Intra-Articular
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — (4-amino-5-(4-(4-(2,4-dichloro-3-(2,4-dimethyl-8-quinolyloxymethyl)phenylsulfonamido)tetrahydro-2H-4-pyranoylcarbonyl)piperazino)-5-oxopentyl)(trimethyl)ammonium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Double dose MEN16132 0.125 mg (Experimental): Intra-articular administration of two 0.125 mg doses of MEN16132 at 2-week interval.
  Interventions: Drug: MEN16132 - 0.125 mg
- Double dose MEN16132 0.25 mg (Experimental): Intra-articular administration of two 0.25 mg doses of MEN16132 at 2-week interval.
  Interventions: Drug: MEN16132 - 0.25 mg
- Double dose MEN16132 0.5 mg (Experimental): Intra-articular administration of two 0.5 mg doses of MEN16132 at 2-week interval.
  Interventions: Drug: MEN16132 - 0.5 mg
- Single dose MEN16132 0.5 mg (Experimental): Intra-articular administration of one 0.5 mg dose of MEN16132 followed by one intra-articular injection of placebo at 2-week interval.
  Interventions: Drug: MEN16132 - 0.5 mg
- Placebo (Placebo Comparator): Intra-articular administration of two doses of Placebo at 2-week interval.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEN16132 - 0.125 mg — Intra-articular administration of two low doses of MEN16132 at 2-week interval.
  Other Names: fasitibant 0.125 mg
  Arms: Double dose MEN16132 0.125 mg
Drug: MEN16132 - 0.25 mg — Intra-articular injection of two intermediate doses of MEN16132 at 2-week interval
  Other Names: fasitibant 0.25 mg
  Arms: Double dose MEN16132 0.25 mg
Drug: MEN16132 - 0.5 mg — Intra-articular injection of two high doses of MEN16132 at 2-week interval
  Other Names: fasitibant 0.5 mg
  Arms: Double dose MEN16132 0.5 mg
Drug: MEN16132 - 0.5 mg — Single intra-articular injection of one high dose of MEN16132, followed by one dose of placebo at 2-week interval
  Other Names: fasitibant 0.5 mg
  Arms: Single dose MEN16132 0.5 mg
Drug: Placebo — Intra-articular injection of 2 doses of Placebo control at 2-week interval
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether intra-articular (knee joint) administration of MEN16132 is effective reducing the pain from knee osteoarthritis.

DETAILED DESCRIPTION:
MEN16132 is a non-peptide bradykinin B2-receptor antagonist showing analgesic and anti-inflammatory activity in nonclinical osteoarthritis models. This study is being conducted as a dose finding study to determine the safety and efficacy of MEN16132, given as three doses/four treatment regimens in comparison to placebo, as well the time to onset and duration of effect.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients ≥40 years old.
* Symptomatic primary knee osteoarthritis (ACR criteria) since ≥6 months prior to screening, Kellgren Lawrence Grade 2 or 3, and representing an indication for intra-articular drug injection.
* >50 mm VAS pain score assigned to the index knee at WOMAC VA 3.1-A1 (pain while walking on a flat surface).
* >125 mm VAS pain score assigned to the index knee at WOMAC VA 3.1 A subscore (total pain).
* Pain in the index knee on at least 50% of the days in the month preceding the screening.

Main Exclusion Criteria:

* Patients with Kellgren & Lawrence Grade I or IV (doubtful or severe) osteoarthritis of the knee.
* Knee condition representing an indication for surgery
* Patients with Inflammatory or crystal arthropathies, acute fractures, severe loss of bone density, bone necrosis.
* Patients with isolated patella-femoral syndrome or chondromalacia.
* Patients with OA predominant in the lateral compartment or any significant valgus deformity.
* Patients with any other disease or condition interfering with the free use and evaluation of the index knee for the 3 month duration of the trial (e.g. cancer, congenital defects, spine osteoarthritis).
* Major injury or surgery to the index knee within the previous 12 months prior to screening.
* Severe hip osteoarthritis ipsilateral to index knee.
* Any pain >30 mm VAS that could interfere with the assessment of index knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee).
* Any pharmacological or non-pharmacological treatment started or changed during 4 weeks prior to randomisation or likely to be changed during the duration of the study
* Use of systemic or topical corticosteroids >10 mg prednisolone equivalent per day during 30 days prior to randomisation.
* Use of any pain or OA medication (e.g. NSAIDs, COX-2 inhibitors, analgesics) during 1 or 2 weeks prior to randomisation.
* Any intra-articular or local periarticular punction, injection or surgery to the index knee during the 6 months prior to screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Pavelka, Prof MD, Principal Investigator — Institute of Rheumatology, Charles University Prague
Locations (23):
- France (3):
  - Centre Hospitalier Régional - Hôpital Porte Madeleine, Orléans
  - Hôtel Dieu - GHU Ouest, Paris
  - Department of Rheumatology, Purpan University Hospital, Toulouse
- Germany (12):
  - Rheumatologie/Immunologie - Rheumazentrum, Krankenhaus Doberan, Bad Doberan
  - Klinik für Rheumatologie und Klinische Immunologie, Charité - Campus Charité Mitte, Berlin
  - Orthopädische Praxis Dr. Wagenitz, Berlin
  - ClinPharm International, Prüfzentrum Bochum, Bochum
  - ClinPharm International, Prüfzentrum Dresden, Dresden
  - Medizinische Klinik 3, Universität Erlangen-Nürnberg, Erlangen
  - ClinPharm Prüfzentrum Frankfurt / aM, Frankfurt
  - ClinPharm Prüfzentrum Görlitz, Görlitz
  - Clinical Research Hamburg, Hamburg
  - Orthopädie Zentrum Altona, Hamburg
  - ClinPharm International, Prüfzentrum Leipzig, Leipzig
  - ClinPharm Prüfzentrum Magdeburg, Magdeburg
- Italy (4):
  - Servizio di Reumatologia, Ospedale Privato Accreditato Nigrisoli, Bologna
  - Dipartimento di Biomedicina - SOD Reumatologia - Azienda Ospedaliera Universitaria Careggi, Florence
  - Dipartimento di Medicina Interna Azienda Ospedaliero Universitaria Pisana-Stabilimento di Santa Chiara Pisa, Pisa
  - Istituto di Reumatologia, "Policlinico Le Scotte" Università degli Studi di Siena, Siena
- Spain (4):
  - Servicio de Reumatologia, Hospital de Basurto, Bilbao
  - Servicio de Reumatologia, Hospital Universitario La Paz, Madrid
  - Servicio de Reumatologia, Corporacio Sanitaria Parc Tauli, Hospital de Sabadell, Sabadell
  - Servicio de Reumatologia, Hospital Universitario Virgen Macarena, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients were recruited from March 2010 to November 2010 in private practice and hospitals.
Groups:
- Low Dose: two intra-articular fasitibant doses; 0.125 mg each
- Mid Dose: two intra-articular fasitibant doses; 0.25 mg each
- High Dose: two intra-articular fasitibant doses; 0.5 mg each
- Single High Dose: one intra-articular fasitibant dose 0.5 mg +placebo
- Placebo: two intra-articular placebo doses
Period: Overall Study
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Started | 83 | 88 | 84 | 84 | 84
Completed | 77 | 80 | 73 | 80 | 73
Not Completed | 6 | 8 | 11 | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Low Dose; Mid Dose; High Dose; Placebo: two doses
- Single High Dose: one dose+placebo
- Total: Total of all reporting groups
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo | Total
Number analyzed (Participants) | 83 | 88 | 84 | 84 | 84 | 423
Age Continuous [Mean (Standard Deviation); unit: years] | 66.7 (9.0) | 65.9 (9.5) | 65.1 (9.7) | 65.3 (8.7) | 65.1 (8.5) | 65.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 51 | 56 | 55 | 252
  Male | 39 | 42 | 33 | 28 | 29 | 171
Duration of osteoarthritis symptoms [Mean (Standard Deviation); unit: years] | 9.7 (9.2) | 8.0 (6.3) | 7.9 (6.6) | 8.2 (8.4) | 6.5 (6.4) | 8.0 (7.5)
Radiographic Osteoarthritis severity [Number; unit: participants] — Based on Kellgren & Lawrence radiologic scale criteria (Grade 1 to 4):
  * narrowing of joint space
  * osteophytic stuctures
  * sclerosis
  * deformity of bone contour
  participants
    Grade 1 Kellgren-Lawrence scale(doubtful severity) | 0 | 0 | 0 | 0 | 0 | 0
    Grade 2 Kellgren-Lawrence scale(minimal severity) | 52 | 45 | 44 | 41 | 42 | 224
    Grade 3 Kellgren-Lawrence scale(moderate severity) | 31 | 43 | 40 | 42 | 42 | 198
    Grade 4 Kellgren-Lawrence scale(severe) | 0 | 0 | 0 | 0 | 0 | 0
    missing information | 0 | 0 | 0 | 1 | 0 | 1
WOMAC VA 3.1 A score (Total pain) [Mean (Standard Deviation); unit: mm] — Western Ontario and McMaster Universities osteoarthritis index (WOMAC). The WOMAC VA 3.1 A score (total pain, range 0-500 mm) is the sum of VAS subscores (0-100 mm) attributed by the patient to each of the 5 questions referring to osteoarthritic pain experienced during the preceding 48 hours (pain domain).
  The higher is the WOMAC VA 3.1 A score, the higher is the intensity of pain symptoms (0 = no pain ; 500 = extreme pain).
  A decrease of the WOMAC VA 3.1 A score following tratment administration indicates a reduction of pain symptom.
  mm | 288 (80) | 282 (68) | 293 (73) | 283 (72) | 284 (79) | 286 (74)

OUTCOME MEASURES:

1. Primary Outcome: WOMAC VA 3.1 A Score (Total Pain)
Description: Western Ontario and McMaster Universities osteoarthritis index (WOMAC). The WOMAC VA 3.1 A score (total pain , range 0-500 mm) is the sum of VAS scores (0-100 mm) attributed by the patient to each of the 5 questions referring to osteoarthritic pain experienced during the preceding 48 hours.
  The higher is the WOMAC VA 3.1 A score, the higher is the intensity of pain symptoms (0 = no pain ; 500 = extreme pain).
  A decrease of the WOMAC VA 3.1 A score following treatment administration indicates a reduction of pain symptom.
  The change from baseline was assessed along 3 weeks after first drug administrations.
Time Frame: over the 3 weeks after the first administration
Population: analysis of the intention to treat (ITT) population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 83 | 88 | 83 | 83 | 84
mm
  1 week post dose 1 | -60 (84) | -58 (82) | -52 (92) | -67 (91) | -63 (103)
  2 weeks post dose 1 | -69 (89) | -65 (81) | -71 (102) | -73 (96) | -75 (93)
  3 weeks post dose 1 | -103 (107) | -99 (86) | -99 (104) | -103 (99) | -103 (112)
Statistical Analysis 1: Comparison: Low Dose vs Mid Dose vs High Dose vs Single High Dose vs Placebo; Tests of Fixed Effects for the primary efficacy variable including baseline treatment and visit (from Visit 3 to Visit 5) as covariates; Test type: Superiority or Other; p = 0.5263, ANCOVA

2. Secondary Outcome: WOMAC VA 3.1.B Score (Knee Stiffness)
Description: WOMAC VA 3.1.B score(range 0-200) is the sum of VAS scores (0-100 mm)attributed by the patient to each of the 2 questions referring to joint stiffness experienced during the preceding 48 hours. The higher is the WOMAC VA 3.1 B score, the higher is joint stiffness (0 = no stiffness ; 200 = extreme stiffness).
  A decrease of the WOMAC VA 3.1 B score following treatment administration indicates a reduction of joint stiffness.
  The change at Week 13 from baseline is reported.
Time Frame: up to 3 months after first dose
Population: Intention to Treat (ITT) population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 83 | 87 | 84 | 83 | 84
mm
  Baseline | 105.7 (47.36) | 101.8 (39.70) | 109.4 (46.21) | 107.3 (43.30) | 108.7 (47.67)
  Week 13 | 61.5 (52.2) | 66.1 (47.4) | 64.5 (50.1) | 66.2 (49.3) | 63.4 (51.3)

3. Secondary Outcome: WOMAC VA 3.1. C Score (Function)
Description: Knee function evaluated by WOMAC VA 3.1 C score (range 0-1700) is the sum of VAS scores (range 0-100 mm) attributed by the patient to each of 17 questions referring to difficulty in performing daily activities experienced during the preceding 48 hours.
  The higher is the WOMAC VA 3.1 C score, the higher is functional impairment in daily activities (0 = no difficulty ; 1700 = extreme difficulty).
  A decrease of the WOMAC VA 3.1 C score following treatment administration indicates an improvement in performing daily activities.
  WOMAC VA 3.1.C scores at baseline and at Week 13 are reported.
Time Frame: up to 3 months after first dose
Population: Intention to Treat (ITT) population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 82 | 88 | 83 | 82 | 83
mm
  Baseline | 928.7 (336.20) | 915.5 (285.20) | 906.7 (318.19) | 938.7 (300.63) | 936.5 (343.80)
  Week 13 | 537.5 (415.9) | 598.0 (396.9) | 574.6 (407.0) | 594.8 (444.3) | 557.6 (389.0)

4. Secondary Outcome: Percentage of Treatment Responders According to OMERACT-OARSI Responder Criteria
Description: Osteoarthritis Research Society International (OARSI).
  Response defined as:
  * a decrease in WOMAC pain or physical-function score by 50% or more and by 20 or more points on the visual analogue scale
  * OR if two of the following three findings are recorded:
  a decrease in the WOMAC pain score by 20% or more and by 10 or more points on the visual analogue scale; a decrease in the WOMAC physical-function score by 20% or more and by 10 or more points on the scale; an improvement in the score on the patient's global assessment by 20% or more and by 10 or more points on the scale.
Time Frame: up to 3 months after first dose
Population: intention to treat (ITT) population
Measure: Number; unit: percentage of patients
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 83 | 88 | 83 | 83 | 84
percentage of patients
  Week 1 | 44.6 | 35.6 | 36.6 | 41.5 | 44.4
  Week 2 | 46.3 | 36.0 | 37.0 | 47.6 | 53.8
  Week 3 | 61.8 | 67.5 | 54.4 | 57.3 | 57.7
  Week 13 | 64.2 | 66.7 | 59.8 | 64.6 | 53.6

5. Secondary Outcome: Patient Global Assessment
Description: Patient global assessment evaluated using a VAS scale score attributed by the patient (range 0-100 mm).
  Efficacy assessed as change at each time-point post-dosing (week 1, 2 ,3, 13) versus baseline (week 0).
  A decrease of patient global assessment score indicates an improvement of osteoarthritis symptoms.
Time Frame: up to 3 months after first dose
Population: intention to treat (ITT) population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 83 | 88 | 83 | 83 | 84
mm
  Week 1 | -4.2 (21.8) | -3.3 (20.4) | 0.9 (18.5) | -6.3 (23.6) | -7.8 (22.2)
  Week 2 | -4.7 (19.6) | -0.4 (21.4) | -0.3 (20.6) | -7.4 (21.9) | -9.0 (24.6)
  Week 3 | -8.4 (25.3) | -4.6 (21.3) | -6.4 (21.5) | -10.2 (24.7) | -11.7 (24.0)
  Week 13 | -14.8 (26.4) | -7.5 (22.3) | -8.8 (23.6) | -11.4 (22.9) | -16.3 (28.8)

6. Secondary Outcome: WOMAC VA 3.1A - Total Pain Score by Body Mass Index [BMI <= 25]
Description: Analysis in normal-weight population (BMI <= 25) of the WOMAC VA 3.1A score (range 0-500 mm) is reported.
  A decrease of the WOMAC VA 3.1 A score following treatment administration indicates a reduction of pain symptom.
Time Frame: over the 3 weeks after the first administration
Population: Population of Normal Weight patients (BMI <=25)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 9 | 15 | 6 | 9 | 12
mm
  1 week post dose 1 | -11.4 (53.91) | -72.4 (55.78) | -109.0 (91.97) | -109.0 (86.66) | 2.7 (75.21)
  2 weeks post dose 1 | 9.2 (97.88) | -90.7 (70.94) | -99.2 (39.89) | -63.8 (90.05) | -31.2 (71.80)
  3 weeks post dose 1 | -22.4 (100.02) | -110.7 (80.72) | -107.8 (46.16) | -112.9 (93.52) | -62.3 (83.43)

7. Secondary Outcome: WOMAC VA 3.1A - Total Pain Score by Body Mass Index -[BMI > 25]
Description: Analysis in over-weight population (BMI > 25) of the WOMAC VA 3.1A score (range 0-500 mm) is reported.
  A decrease of the WOMAC VA 3.1 A score following treatment administration indicates a reduction of pain symptom.
Time Frame: over the 3 weeks after the first administration
Population: Population of Over Weight patients (BMI >25)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 29 | 36 | 38 | 30 | 28
mm
  1 week post dose 1 | -76.5 (81.73) | -62.9 (81.14) | -56.4 (88.08) | -67.4 (86.99) | -58.0 (70.92)
  2 weeks post dose 1 | -88.2 (83.18) | -78.2 (75.67) | -81.5 (105.08) | -81.6 (90.11) | -83.9 (72.71)
  3 weeks post dose 1 | -103.4 (95.60) | -122.1 (69.96) | -114.1 (106.00) | -99.6 (83.74) | -103.3 (85.26)

8. Secondary Outcome: Adverse Event Reports
Description: Incidence of spontaneously reported adverse events
Time Frame: up to 4 months after screening
Population: The number of patients reflects all patients administered at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 83 | 88 | 83 | 83 | 84
participants
  Non-serious adverse events | 31 | 38 | 36 | 28 | 33
  Serious adverse events | 1 | 2 | 3 | 3 | 2
  Blood / Lymph system | 0 | 0 | 0 | 1 | 0
  Cardiac disorders | 2 | 3 | 1 | 2 | 1
  Eye disorders | 0 | 0 | 0 | 1 | 0
  Gastrointestinal disorders | 5 | 3 | 2 | 2 | 2
  General / administration site conditions | 3 | 4 | 6 | 3 | 3
  Infections / infestations | 11 | 11 | 10 | 10 | 10
  Injury / poisoning / procedural complications | 3 | 4 | 5 | 2 | 3
  Investigations | 2 | 3 | 3 | 2 | 3
  Metabolism and nutrition disorders | 1 | 0 | 0 | 0 | 2
  Musculoskeletal and connective tissue disorders | 6 | 11 | 11 | 10 | 12
  Nervous system disorders | 6 | 3 | 5 | 3 | 3
  Psychiatric disorders | 1 | 0 | 2 | 0 | 0
  Renal and Urinary disorders | 0 | 0 | 0 | 0 | 2
  Respiratory, thoracic, and mediastinal disorders | 0 | 1 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders | 1 | 0 | 1 | 1 | 1
  Surgical and medical procedures | 1 | 0 | 1 | 1 | 1
  Vascular disorders | 4 | 4 | 2 | 4 | 2
  Social circumstances | 0 | 1 | 0 | 0 | 0

9. Secondary Outcome: Clinically Significant Abnormal Laboratory Tests
Description: Percentage of patients with Abnormal Laboratory Tests judged Clinically Significant by Investigators.
  The following hematochemical and urinary parameters were analysed:
  Red Blood Cells Count, Haematocrit, Haemoglobin, Platelets, MCV, MCH, MCHC, White Blood Cells, Sodium, Chloride, Potassium, Total calcium, AST (SGOT), ALT (SGPT), GGT, Alkaline phosphatase, Total Bilirubin, Direct Bilirubin, Creatinine, BUN, CPK, LDH, Glucose, Total proteins, Albumin.
Time Frame: up to 4 months from screening
Population: Percentage of patients with clinically significant abnormal laboratory tests
Measure: Number; unit: participants
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Number analyzed (Participants) | 83 | 88 | 84 | 84 | 84
participants
  Blood GGT | 0 | 0 | 1 | 0 | 1
  Blood Alkaline Phophatase | 0 | 0 | 1 | 0 | 0
  Blood Total Bilirubin | 0 | 0 | 1 | 0 | 0
  Blood Creatinine | 0 | 1 | 0 | 0 | 0
  Blood Glucose | 0 | 0 | 0 | 1 | 1
  Blood Potassium | 0 | 0 | 1 | 0 | 1
  Blood Sodium | 0 | 0 | 0 | 0 | 1
  Blood Fibrin D dimer | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Four months of safety observation
Arm/Group | Low Dose | Mid Dose | High Dose | Single High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 1/83 | 2/88 | 3/83 | 3/83 | 2/84
Other Adverse Events (participants affected / at risk) | 17/83 | 18/88 | 21/83 | 15/83 | 16/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=83) | Mid Dose (N=88) | High Dose (N=83) | Single High Dose (N=83) | Placebo (N=84)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular-tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain Barré syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uretric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterocele (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=83) | Mid Dose (N=88) | High Dose (N=83) | Single High Dose (N=83) | Placebo (N=84)
Injection site pain (General disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5) | 4 (4) | 4 (5) | 5 (6)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (5) | 7 (7) | 6 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No